CLINICAL TRIAL: NCT04293926
Title: Effects of a Resistance Training Program on Heart Rate Variability in Children and Adolescents With Cystic Fibrosis
Brief Title: Heart Rate Variability in Children and Adolescents With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Margarita Perez, Full Professor In Exercise Physiology, MD, PhD, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UEM50
Record Dates: First submitted 2020-02-25; First posted 2020-03-03 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Cystic Fibrosis in Children
Keywords: Cystic Fibrosis; Heart Rate Variability; Exercise
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This group will receive routine recommendations by the pediatrician, including specific lifestyle advises.
- Exercise (Experimental): This group will receive routine recommendations by the pediatrician, including specific lifestyle advises. In addition, a 8-week resistance exercise training program will be performed.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Resistance exercise program for 8 weeks, 3 times a week, with a 60 min session duration.
  Arms: Exercise

SUMMARY:
This study aims to assess the effects of a resistance exercise training program on heart rate variability in a group of children and adolescents with cystic fibrosis. The study design is a randomized controlled trial.

DETAILED DESCRIPTION:
A randomized controlled study will be carried out in children diagnosed with cystic fibrosis aged 6 to 18 years. Individuals will be divided into two groups: control group (CON) and strength training (ST). Heart rate variability will be analyzed using KUBIOS and measured using a Suunto watch, with subjects in lying position without movements or speaking for 5 minutes. Patients in the ST group will complete an individualized guided strength program for 8 weeks (3 sessions of 60 min/week). Training prescription will be individualized and based on the 5 repetition maximum test (60-80%). Upper and lower limbs exercises will be used, including seated bench press, seated lateral row and leg press. Outcome measures will be performed at baseline and after 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cystic Fibrosis
* Age between 6 and 18 years old
* Mild to moderate lung function levels
* Signature of the informed consent form by legal guardian and patient.

Exclusion Criteria:

* Active smoking
* Exacerbation in the last 3 months
* Presence of gastrostomy
* Use of beta-blocker drugs
* Diagnosed heart disease
* Alterations in the locomotor system

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
Change in the standard deviation of R-R intervals (SDNN) expressed in milliseconds (m/s) | Baseline and 8 weeks
  Changes in time-domain SDNN will be measured through heart rate variability assessment using a heart rate band and an Ambit 3 Sport watch. Variables will be collected during a five minute period.
Change in the root mean square standard deviation (RMSSD) expressed in milliseconds (m/s) | Baseline and 8 weeks
  Changes in time-domain RMSSD will be measured through heart rate variability assessment using a heart rate band and an Ambit 3 Sport watch. Variables will be collected during a five minute period.
Change in the percentage of differences between R-R intervals higher than 50 m/s (PNN50) expressed in percentage (%) | Baseline and 8 weeks
  Changes in time-domain PNN50 will be measured through heart rate variability assessment using a heart rate band and an Ambit 3 Sport watch. Variables will be collected during a five minute period.
Change in the low frequency band (LF) expressed in normalized unites (nu) | Baseline and 8 weeks
  Changes in frequency-domain LF will be measured through heart rate variability assessment using a heart rate band and an Ambit 3 Sport watch. Variables will be collected during a five minute period.
Change in the high frequency band (HF) expressed in normalized unites (nu) | Baseline and 8 weeks
  Changes in frequency-domain HF will be measured through heart rate variability assessment using a heart rate band and an Ambit 3 Sport watch. Variables will be collected during a five minute period.
Change in the quotient (LF/HF) between the low frequency band (LF) and the high frequency band (HF) expressed as a ratio | Baseline and 8 weeks
  Changes in frequency-domain HF will be measured through heart rate variability assessment using a heart rate band and an Ambit 3 Sport watch. Variables will be collected during a five minute period.

SECONDARY OUTCOMES:
Change in the forced expiratory volume in one second (FEV1) expressed as z-score | Baseline and 8 weeks
  Changes in FEV1 will be measured using spirometry
Change in the forced vital capacity (FVC) expressed as z-score | Baseline and 8 weeks
  Changes in FVC will be measured using spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Perez Ruiz, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Escuela de Doctorado e Investigacion, Universidad Europea, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Estevez-Gonzalez AJ, Donadio MVF, Cobo-Vicente F, Fernandez-Luna A, Sanz-Santiago V, Villa Asensi JR, Iturriaga Ramirez T, Fernandez-Del-Valle M, Diez-Vega I, Larumbe-Zabala E, Perez-Ruiz M. Effects of a Short-Term Resistance-Training Program on Heart Rate Variability in Children With Cystic Fibrosis-A Randomized Controlled Trial. Front Physiol. 2021 Mar 30;12:652029. doi: 10.3389/fphys.2021.652029. eCollection 2021. PMID 33859572